CLINICAL TRIAL: NCT00745407
Title: Effects of Fenofibrate on Adipocytokine Levels In Hypertriglyceridemic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Model: Crossover | Purpose: Treatment
Other Study IDs: GMC 200511
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Hypertriglyceridemia
Keywords: adipocytokines; insulin sensitivity; hypertriglyceridemic patients
MeSH Terms: conditions — Hypertriglyceridemia; Insulin Resistance | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fenofibrate 160 mg, placebo (Experimental)
  Interventions: Drug: fenofibrate

INTERVENTIONS:
Drug: fenofibrate

SUMMARY:
Fenofibrate increases adiponectin levels, but reduces leptin levels

ELIGIBILITY:
Inclusion Criteria:

* hypertriglyceridemia

Exclusion Criteria:

* chronic liver disease

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea